CLINICAL TRIAL: NCT07282613
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) s.c. Once Weekly Versus Placebo in Children and Adolescents With Type 2 Diabetes
Brief Title: A Research Study to See How Much CagriSema Lowers Blood Sugar and Body Weight Compared to Placebo in Children and Adolescents With Type 2 Diabetes
Acronym: REIMAGINEYOUNG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-7988; U1111-1307-6786 (Other: World Health Organization (WHO)); 2024-514432-24 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: It is 2-part study, first part is double-blinded and second part is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: CagriSema (Experimental): Participants will receive CagriSema (Cagrilintide B + Semaglutide I) subcutaneously once weekly for 26 weeks in Part 1.
  Interventions: Drug: CagriSema (Cagrilintide B and Semaglutide I)
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo matched to CagriSema (Cagrilintide B + Semaglutide I) subcutaneously once weekly for 26 weeks in Part 1.
  Interventions: Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I)
- Part 2: CagriSema (Experimental): Participants who received placebo in Part 1 will receive CagriSema (Cagrilintide B + Semaglutide I) subcutaneously once weekly for 26 weeks in Part 2.
  Interventions: Drug: CagriSema (Cagrilintide B and Semaglutide I)

INTERVENTIONS:
Drug: CagriSema (Cagrilintide B and Semaglutide I) — Cagrilintide B and Semaglutide I will be administered subcutaneously using DV3384 pen-injector.
  Arms: Part 1: CagriSema; Part 2: CagriSema
Drug: Placebo matched to CagriSema (Cagrilintide B and Semaglutide I) — Placebo matched to Cagrilintide B and Placebo matched to Semaglutide I will be administered subcutaneously using DV3384 pen-injector.
  Arms: Part 1: Placebo

SUMMARY:
The purpose of this clinical study is to look into how well a study medicine called CagriSema helps children and adolescents living with diabetes lower their blood sugar and body weight. The study has 2 parts: in the first part participant will get either CagriSema or placebo, and in the second part participant will get CagriSema. In the first part, which treatment participant gets is decided by chance and second part is open label and all participants will get CagriSema during this part. The study will last for about 1 year and 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent of parent(s) or legally acceptable representative (LAR) of participant and child assent, as age-appropriate, obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.

  * The parent(s) or LAR of the child must sign and date the Informed Consent Form (according to local requirements)
  * The child must sign and date the Child Assent Form or provide oral assent (according to local requirements)
* Male or female.
* Age 10 to < 18 years at the time of signing the informed consent.
* Diagnosed with T2D (according to the latest International Society for Pediatric and Adolescent Diabetes [ISPAD] criteria) ≥ 30 days before screening.
* Treated with diet and exercise counselling alone or with a stable daily dose(a), in addition to diet and exercise counselling, of any of the following antidiabetic drugs or combination regimens:

  * Insulin (any regimen)
  * Metformin
  * SGLT2i
* HbA1c 6.5%-11.0% (48 mmol/mol - 97 mmol/mol) (both inclusive) as determined by central laboratory at screening.
* Body weight ≥ 45 kg and BMI ≥ 85th percentile(b). BMI will be calculated in the electronic case report form based on height and body weight at screening.

  * (a) For metformin, a stable dose is defined as at least 1000 mg daily or the maximum tolerated dose for ≥ 56 days prior to screening. For Sodium-Glucose Transport protein 2 inhibitor (SGLT2i), a stable dose is defined as the same total daily dose for ≥ 56 days prior to screening. For insulin, it is defined as the dose ± 25% of that taken at screening for ≥ 30 days prior to screening.
  * (b) Based on sex-specific BMI-for-age percentiles for the given country or region. If not available for the country or region, the respective charts or tables on cdc.gov may be used.

Key Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Treatment with any antidiabetic or anti-obesity medication (irrespective of indication) other than stated in the inclusion criteria within 90 days before screening.
* Known or previous diagnosis of hypoparathyroidism.
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device. However, the following are allowed: (1) liposuction and/or abdominoplasty, if performed >1 year before screening, (2) lap banding, if the band has been removed >1 year before screening, (3) intragastric balloon, if the balloon has been removed >1 year before screening or (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening.
* Positive insulinoma associated-protein 2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies as determined by central laboratory at screening or in medical history.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8.
* Uncontrolled and potentially unstable diabetic retinopathy maculopathy. Verified by a fundus examination and optical coherence tomography (OCT) assessment performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-08-04 (Estimated); Primary Completion 2029-09-07 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as percentage (%) of HbA1c.

SECONDARY OUTCOMES:
Relative change in body mass index (BMI) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as percentage.
Number of participants with achievement of HbA1c target values of less than (<) 7.0% (< 53 millimole per mole [mmol/mol]) | At end of double-blinded treatment (week 26)
  Measured as count of participants.
Number of participants with achievement of HbA1c target values of less than or equal to (≤) 6.5% (≤48 mmol/mol) | At end of double-blinded treatment (week 26)
  Measured as count of participants.
Change in time in range (TIR) 3.9-10.0 millimole per liter (mmol/L) (70-180 milligram per deciliter (mg/dL) measured using continuous glucose monitoring (CGM) | From baseline (collected during week -3, -2 and -1) to end-of-double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Change in time in tight target range (TITR) 3.9-7.8 mmol/L (70-140 mg/dL) measured using CGM | From baseline (collected during week -3, -2 and -1) to end-of-double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Change in time above range (TAR) greater than (>) 10.0 mmol/L (> 180 mg/dL) measured using CGM | From baseline (collected during week -3, -2 and -1) to end-of-double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Change in TAR greater than (>) 13.9 mmol/L (> 250 mg/dL) measured using CGM | From baseline (collected during week -3, -2 and -1) to end-of-double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Change in mean sensor glucose concentration measured by CGM | From baseline (collected during week -3, -2 and -1) to end-of- double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as mmol/L.
CGM: Within-day glycaemic variability (% coefficient of variation) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as percentage.
Number of participants with incidence of glycaemic rescue therapy | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of participants
Change in fasting plasma glucose | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as mmol/L.
Number of participants with achievement of greater than or equal to (≥) 5% BMI reduction | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of participants.
Number of participants with achievement of ≥ 10% BMI reduction | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of participants.
Number of participants with achievement of ≥ 15% BMI reduction | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of participants.
Relative change in body weight | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as percentage of body weight.
Change in BMI standard deviation score (SDS) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as score on scale.
Change in waist circumference | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as centimetre (cm).
Change in waist-to-height ratio | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Change in systolic blood pressure | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as millimetre of mercury (mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as mmHg.
Ratio to baseline in lipid: total cholesterol | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in lipid: high density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in lipid: low density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in lipid: very low density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in lipid: triglycerides | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in lipid: Non-HDL cholesterol | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Change in alanine aminotransferase (ALT) | From baseline (week 0) to end of double-blinded treatment (week 26) and end of extension phase treatment (week 52)
  Measured as units per liter (U/L).
Apparent clearance (CL/F) of cagrilintide and semaglutide | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as liter per hour (L/h).
Average concentration (Cavg) of cagrilintide and semaglutide at steady state | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as nanomole per liter (nmol/L).
Change in insulin dose | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as units (U).
Number of participants with achievement of sustained insulin dose = 0 U | At end of double-blinded treatment (week 26)
  Measured as count of participants.
Ratio to baseline in urine albumin-creatinine ratio (UACR) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in biomarker related to glucose metabolism: fasting C-peptide | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in biomarker related to glucose metabolism: fasting insulin | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in biomarker related to glucose metabolism: fasting proinsulin | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in biomarker related to glucose metabolism: fasting glucagon | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in high sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to end of double- blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in free fatty acids | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in leptin | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in soluble leptin receptor | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Ratio to baseline in leptin to soluble leptin receptor ratio | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as ratio.
Change in aspartate aminotransferase (AST) | From baseline (week 0) to end of double-blinded treatment (week 26) and end of extension phase treatment (week 52)
  Measured as U/L.
Change in alkaline phosphatase (ALP) | From baseline (week 0) to end of double-blinded treatment (week 26) and end of extension phase treatment (week 52)
  Measured as U/L.
Change in bilirubin | From baseline (week 0) to end of double-blinded treatment (week 26) and end of extension phase treatment (week 52)
  Measured as U/L.
Change in HbA1c | From baseline (week 0) to end of extension phase treatment (week 52)
  Measured as percentage of HbA1c.
Number of clinically significant hypoglycaemic episodes (level 2) (< 3.0 mmol/L (54 mg/dL) confirmed by blood glucose [BG] meter) | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of episodes.
Number of severe hypoglycaemic episodes (level 3) - severe hypoglycaemia being defined as severe cognitive impairment requiring assistance by another person to administer carbohydrates, glucagon, or intravenous glucose | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of episodes.
Change in percentage of time below range (TBR) < 3.0 mmol/L (< 54 mg/dL) measured using CGM | At end of double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Change in TBR < 3.9 mmol/L (< 70 mg/dL) measured using CGM | At end of double-blinded treatment (collected during week 22, 23, 24, and 25)
  Measured as percentage of time.
Number of treatment-emergent adverse events | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as count of events.
Height velocity | At end of double-blinded treatment (week 26)
  Measured as cm/year.
Change in height SDS | From baseline (week 0) to end of double-blinded treatment (week 26)
  Measured as score on scale.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (54):
- United States (20):
  - Yale School of Medicine, New Haven, Connecticut
  - Encore Medical Research Boynton Beach, Boynton Beach, Florida
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Innovus Clinical, Kissimmee, Florida
  - D&H National Research Centers, Tamarac, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - Columbus Research Foundation, Columbus, Georgia
  - Eastside Bariatric and Gen Surg, Snellville, Georgia
  - SIU Medicine, Springfield, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Great Lakes Research Inst., Southfield, Michigan
  - UBMD Pediatrics, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - LifeDoc Health, Memphis, Tennessee
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Seattle Children's Research Institute, Seattle, Washington
- Argentina (4):
  - Centro de Investigación C.I.C.E 9 de Julio - Sanatorio 9 de Julio, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Metabólicas, Capital Federal
  - IMOBA, City of Buenos Aires
  - Clínica Mayo de Urgencias Médicas Cruz Blanca, San Miguel de Tucumán
- Brazil (5):
  - Hospital Universitário Walter Cantídio, Bairro Rodolfo Teófilo, Fortaleza, Ceará
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Instituto da Criança com Diabetes - ICD, Porto Alegre, Rio Grande do Sul
  - Unidade de Pesquisa Clínica do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Instituto da Criança e do Adolescente do HCFMUSP, São Paulo, São Paulo
- Colombia (2):
  - Salud SURA Industriales, Bogotá, Antioquia
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
- India (9):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - Indira Gandhi Institute of child health, Bangalore, Karnataka
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Maulana Azad Medical College, Delhi, New Delhi
  - Regency Hospital, Kanpur, Uttar Pradesh
  - Institute of Child Health, Kolkata, West Bengal
  - Excel Endocrine Centre, Kolhāpur
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Israel (5):
  - HaEmek MC - Pediatric Endocrinology department, Afula
  - Soroka MC - Pediatric Endocrinology, Beersheba
  - Rambam MC - Department of Pediatrics A, Haifa
  - Carmel MC - Pediatric Endocrinology Unit, Haifa
  - Shaare Zedek MC - Pediatric Endocrinology, Jerusalem
- Malaysia (2):
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya
- Mexico (4):
  - Instituto Nacional de Pediatría, Coyoacán, Mexico City
  - IECSI Centro de Investigación Clínica, Monterrey, Nuevo León
  - Centro de Investigación y Control Metabólico S. C., San Nicolás de los Garza, Nuevo León
  - Consultorio de Endocrinología y Pediatría, Puebla City
- Taipei Mackay Memorial Hospital, Taipei, Taiwan
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital_Pediatric Endocrinology, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com